CLINICAL TRIAL: NCT05878158
Title: Clinical and Digital Radiographic Evaluation of Simvastatin Versus MTA in Pulpotomy of Immature Permanent Vital Molars: A18 Month Randomized Controlled Trial
Brief Title: Simvastatin Versus MTA in Pulpotomy of Immature Permanent Molars
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmad Elheeny (Other)
Responsible Party: Sponsor-Investigator, Ahmad Elheeny, clinical professor, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300
Record Dates: First submitted 2023-05-02; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Pulp Exposure, Dental
MeSH Terms: conditions — Dental Pulp Exposure | interventions — Simvastatin; mineral trioxide aggregate

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simvastatin (Active Comparator): Drug The drug powder will be mixed with distilled water to form a paste applied in the pup chamber of immature permanent molars over the pulp stump
  Interventions: Drug: Simvastatin
- Mineral Trioxide Aggregate (Experimental): Dental material It is a regenrative endodontic material prepared as apoweder that mixed with distilled water to form a paste applied in the pup chamber of immature permanent molars over the pulp stump
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — pulpotomy of immature permanent teeth
  Other Names: Mineral Trioxide Aggregate

SUMMARY:
the study will be done to evaluate the clinical and digital radiographic success of simvastatin versus MTA in pulpotomy of immature permanent molars

DETAILED DESCRIPTION:
the clinical and digital radiographic success of simvastatin versus MTA in pulpotomy of immature permanent molars for the following patients which include: Healthy children aged from 6 to 8 years who will be classified as Class I or II Children according to the American Society of Anaesthesiologists (ASA) will be included. Children with severe behavioral, or emotional disabilities, and medically compromised children will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged from 6 to 8 years
* Children with severe behavioral, or emotional disabilities, and medically compromised children will be excluded.
* Deep carious lesions of the first permanent immature molars with signs & symptoms of reversible pulpitis will be included
* Normal radiographic findings and immature roots

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of pain | one year
  clinical assessment

SECONDARY OUTCOMES:
Dentin wall thickness | 18 months
  radiographic assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided